CLINICAL TRIAL: NCT04418583
Title: Quantifying the Effect of the Crane Technique Through Three-dimensional Imaging
Acronym: CRANE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: METCZ20200071
Record Dates: First submitted 2020-05-20; First posted 2020-06-05 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-05

CONDITIONS: Pectus Excavatum; Funnel Chest
MeSH Terms: conditions — Funnel Chest | interventions — Imaging, Three-Dimensional

STUDY DESIGN:
Intervention Model Description: Prospective case-control study wherein participants are their own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three-dimensional imaging (Experimental): Participants receive a three-dimensional image of their chest, just prior to and after application of the Crane technique.
  Interventions: Diagnostic Test: Three-dimensional imaging

INTERVENTIONS:
Diagnostic Test: Three-dimensional imaging — Three-dimensional surface images, acquired by the Artec Leo

SUMMARY:
Pectus excavatum is the most common congenital abnormality of the thoracic wall and occurs in 1 in 400 newborns. The gold standard treatment is the Nuss bar Procedure. However, in very severe cases, pectus exacavatum involves little or no space between the heart and sternum. Because of the limited space, the Nuss procedure is more difficult to perform and there is an increased risk of complications such as injuries to the heart or large vessels. However, this increased risk can again be reduced by using the Crane technique. This technique increases the substernal space by sternal 'hoisting' via an external steel wire. Despite the fact that this technique is commonly used, it is not known what its quantitative effect is on the substernal space during the Nuss bar procedure. The subsequent aim of this study is to quantify the effect of the Crane technique during minimally invasive repair of pectus excavatum through three-dimensional scans acquired before and after application of the Crane technique.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing minimally invasive repair of pectus excavatum (through the Nuss bar procedure) in conjunction with the Crane technique.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Mean change in chest wall dimensions | 1 hour
  difference between baseline (first image) and image after application of the Crane technique

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Centre, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided